CLINICAL TRIAL: NCT04507958
Title: The Accuracy of Electronic Stethoscope for Confirmation of Endotracheal Intubation Position in Full Personal Protective Equipment
Brief Title: Electronic Stethoscope Use During Intubation in Full Personal Protective Equipment
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005104RINC
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2020-08

CONDITIONS: Thoracic Surgery
Keywords: endotracheal intubation; electronic stethoscope; personal protective equipment

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electronic auscultation
  Interventions: Diagnostic Test: auscultation by using electronic stethoscope in full PPE
- Conventional ausculatation
  Interventions: Diagnostic Test: auscultation by using conventional stethoscope without PPE

INTERVENTIONS:
Diagnostic Test: auscultation by using conventional stethoscope without PPE — In thoracic patients undergoing general anesthesia with endotracheal tube/endobronchial blocker, Clinician will check the position of endotracheal tube and endobronchial blocker under fiberscope. Afterward, investigator A will perform auscultation with traditional auscultation, then investigator B with electronic stethoscope under full PPE, to examine bilateral breathing sound.
  Groups: Conventional ausculatation
Diagnostic Test: auscultation by using electronic stethoscope in full PPE — In thoracic patients undergoing general anesthesia with endotracheal tube/endobronchial blocker, Clinician will check the position of endotracheal tube and endobronchial blocker under fiberscope. Afterward, investigator A will perform auscultation with traditional auscultation, then investigator B with electronic stethoscope under full PPE, to examine bilateral breathing sound.
  Groups: Electronic auscultation

SUMMARY:
To investigate the feasibility of auscultation to confirm the endotracheal tube position by using electronic stethoscope for clinicians who wear the full personal protective equipment.

DETAILED DESCRIPTION:
After the pandemic outbreak of Coronavirus disease 2019 (COVID-19) in many countries, the number of critical ill patients are rapidly growing. Critical ill COVID-19 patients inevitably require endotracheal intubation for ventilator support. The chest X-rays, ultrasound, and stethoscope are three tools that can detect whether or not bronchial intubation has occurred. Auscultation by using the stethoscope is the routine first-line tool for this purpose. However, clinician who wears the full personal protective equipment (PPE) is very difficult to perform adequate auscultation with conventional stethoscope. In addition, the X-ray machines and ultrasound are very difficult to enter the negative-pressure isolation room and may raise the risks of infection spread. By using the electronic stethoscope amplified by the Bluetooth speaker, the clinician with full PPE may still hear the proper lung sound. In addition, electronic stethoscope has a good portability that can be easily brought into the isolation room. For patients undergoing surgery with general anesthesia, endotracheal tube is often mandatory and auscultation with stethoscope is routinely applied. Therefore, the investigators can simulate the circumstance that clinician with a full PPE to use the electronic stethoscope for confirmation of the proper endotracheal tube position. In addition, patients undergoing thoracic surgery require the single-lung ventilation which could be a proper simulation scenario for detection of bronchial intubation by using electronic stethoscope for clinicians with PPE.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery in general anesthesia with endotracheal tube insertion and bronchial blocker.

Exclusion Criteria:

* Previous lung surgical history
* Patients with organs dysfunction, such as impaired liver function, eg. Aspartate Aminotransferase or Alanine Aminotransferase >100; liver cirrhosis > Child B class; impaired renal function, calculated glomerulus filtration rate< 60 ml/min/1.73 m2; cardiac dysfunction, such as heart failure > New York Heart Association class II, coronary arterial disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients meeting the eligibility criteria undergoing thoracic surgery in general anesthesia with endotracheal tube insertion and bronchial blocker will be assessed for informed consent
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
The ability to detect selective lung isolation states | 90 seconds
  Perform the auscultation by investigator A with traditional stethoscope, then by investigator B with electronic stethoscope under full PPE, to detect bronchial or tracheal intubation. The accuracy of successful detection (%) is the primary outcome.

SECONDARY OUTCOMES:
User experience of the electronic stethoscope | Through study completion, an average of 1 year
  After complete of the trial, participant physicians will be asked to report the questionnaire of the experience of using electronic stethoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Taiwan National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsingh D, Frank E, Haughton R, Schilling J, Gimenez KM, Banh E, Rinehart J, Cannesson M. Auscultation versus Point-of-care Ultrasound to Determine Endotracheal versus Bronchial Intubation: A Diagnostic Accuracy Study. Anesthesiology. 2016 May;124(5):1012-20. doi: 10.1097/ALN.0000000000001073. PMID 26950708